CLINICAL TRIAL: NCT04822077
Title: PROTHYM - Phase II Non-randomized Study on Proton Radiotherapy Of Thymic Malignancies
Brief Title: Study on Proton Radiotherapy of Thymic Malignancies
Acronym: PROTHYM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ass. Prof. Jan Nyman (Network)
Responsible Party: Sponsor-Investigator, Ass. Prof. Jan Nyman, Head of Swedish Lung Cancer Study Group, Ass. Prof., Swedish Lung Cancer Study Group
Organization: Swedish Lung Cancer Study Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROTHYM 2.2
Record Dates: First submitted 2021-03-11; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Cardiotoxicity; Pulmonary Toxicity; Thymus Neoplasms
Keywords: Thymoma; Thymic carcinoma; Proton radiotherapy
MeSH Terms: conditions — Cardiotoxicity; Thymus Neoplasms; Thymoma | interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: Phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton radiotherapy (Experimental): Proton radiotherapy with RBE doses:
  * Patients with radical surgery and unfavourable histology (B2, B3, C) and/or Masaoka-Koga stage III, IVa: 2 Gy(RBE), once daily, five days a week to a total dose of 50 Gy(RBE).
  * Patients with non-radical surgery (R1 resection) regardless of stage and histology: 2.3 Gy(RBE), once daily, 5 days a week to a total dose of 57.5 Gy(RBE)
  * Inoperable patients regardless of stage and histology and patients with R2 non-radical resection: 2.5 Gy (RBE), once daily, 5 days a week to a total dose of 62.5 Gy(RBE)
  Interventions: Radiation: Proton radiation

INTERVENTIONS:
Radiation: Proton radiation — * Patients with radical surgery and unfavourable histology (B2, B3, C) and/or Masaoka-Koga stage III, IVa: 2 Gy(RBE), once daily, five days a week to a total dose of 50 Gy(RBE).
  * Patients with non-radical surgery (R1 resection) regardless of stage and histology: 2.3 Gy(RBE), once daily, 5 days a week to a total dose of 57.5 Gy(RBE)
  * Inoperable patients regardless of stage and histology and patients with R2 non-radical resection: 2.5 Gy (RBE), once daily, 5 days a week to a total dose of 62.5 Gy(RBE)

SUMMARY:
This is a multicentre non-randomized phase II study of proton beam radiotherapy in patients with thymic epithelial tumours (i.e. thymoma and thymic carcinoma) in the post-operative setting or in inoperable patients with localized disease.

Patients not willing or for any reason unsuitable to undergo proton treatment will be asked to participate in a follow-up assessment after the regular photon treatment in the same manner as the included patients.

Primary endpoints are:Toxicity (e.g. cardiac and pulmonary toxicity) and Local control at 5 year Secondary endpoints: PFS, Overall survival, Quality of life, measured by EORTC QLQ 30 + LC 13 and relapse pattern

DETAILED DESCRIPTION:
All doses are recorded in Gy(RBE).

After having checked all eligibility criteria patients will receive:

* Patients with radical surgery and unfavourable histology (B2, B3, C) and/or Masaoka-Koga stage III, IVa: 2 Gy(RBE), once daily, five days a week to a total dose of 50 Gy(RBE).
* Patients with non-radical surgery (R1 resection) regardless of stage and histology: 2.3 Gy(RBE), once daily, 5 days a week to a total dose of 57.5 Gy(RBE)
* Inoperable patients regardless of stage and histology and patients with R2 non-radical resection: 2.5 Gy (RBE), once daily, 5 days a week to a total dose of 62.5 Gy(RBE)
* Patients not willing to participate in study will receive photon therapy according to local practice (≥45 Gy)

Induction or adjuvant chemotherapy may be used according to local practice. Concomitant chemotherapy is not allowed.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of thymoma or thymic carcinoma.
* With radical surgery: stage III and IVa and selected stage II with type B2, B3 and thymic carcinoma according to local routine. With non-radical surgery (R1 or R2) or inoperable patient/ patient refusing surgery: stage I - IVa, any histology
* PS WHO 0 - 2.
* FEV1 > 1L or >40 % of predicted and CO diffusion capacity > 40% of predicted (postoperative measures)
* Age >18 years, no upper age limit.
* Written informed consent from patients.

Exclusion Criteria:

* Masaoka-Koga stage IVb (distant metastases).
* Pregnancy.
* Serious concomitant systemic disorder incompatible with the study.
* Tumour motion > 0.5 cm on two repeated 4DCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Cardiotoxicity and pulmonary toxicity of therapy | At 60 months from treatment
  Proportion of patients with cardiac and pulmonary toxicity measured by CTCAE 4.0 > Grade 2
Local tumor control | At 60 months from treatment
  Freedom from tumor progression (CR,PR or SD) mesured by CT-scan

SECONDARY OUTCOMES:
Quality of life questionnaire EORTC QLQ 30 (European Organisation for Research and Treatment of Cancer) | At 60 months from treatment
  Scale from 1-100 for 30 items, higher score indicates a better situation.
Quality of life questionnaire LC13 (Lung cancer specific module of EORTC) | At 60 months from treatment
  Scale from 1-100 for 13 items and higher score indicates worse symptoms.
Survival | From treatment and for 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Hillevi Rylander, MD, Study Director — Head of Skandion Clinic
Locations (3):
- Sweden (3):
  - Department of Oncology, Norrlands Universitetssjukhus, Umeå, Norrland
  - Department of Oncology, Karolinska University Hospital, Stockholm, Stockholm County
  - Department of Oncology, Sahlgrenska University Hospital, Gothenburg, Västra Götaland County

IPD SHARING:
Plan to Share IPD: No
The aim is that the study will be published in international journals. A separate publication will include result of the cardiological data The Vancouver declaration (Br Med J:296, 401-405, 1988) should be followed in all publications based on this study.

REFERENCES:
- [Result] Chang JY, Li H, Zhu XR, Liao Z, Zhao L, Liu A, Li Y, Sahoo N, Poenisch F, Gomez DR, Wu R, Gillin M, Zhang X. Clinical implementation of intensity modulated proton therapy for thoracic malignancies. Int J Radiat Oncol Biol Phys. 2014 Nov 15;90(4):809-18. doi: 10.1016/j.ijrobp.2014.07.045. Epub 2014 Sep 24. PMID 25260491
- [Result] Gomez D, Komaki R. Technical advances of radiation therapy for thymic malignancies. J Thorac Oncol. 2010 Oct;5(10 Suppl 4):S336-43. doi: 10.1097/JTO.0b013e3181f20ea2. PMID 20859129
- [Result] Vogel J, Berman AT, Lin L, Pechet TT, Levin WP, Gabriel P, Khella SL, Singhal S, Kucharczuk JK, Simone CB 2nd. Prospective study of proton beam radiation therapy for adjuvant and definitive treatment of thymoma and thymic carcinoma: Early response and toxicity assessment. Radiother Oncol. 2016 Mar;118(3):504-9. doi: 10.1016/j.radonc.2016.02.003. Epub 2016 Feb 16. PMID 26895711
- [Result] Bjork-Eriksson T, Bjelkengren G, Glimelius B. The potentials of proton beam radiation therapy in malignant lymphoma, thymoma and sarcoma. Acta Oncol. 2005;44(8):913-7. doi: 10.1080/02841860500355983. PMID 16332601

DOCUMENTS (1):
  • Study Protocol (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT04822077/Prot_000.pdf